CLINICAL TRIAL: NCT03363698
Title: The Usefulness of the Methacholine Challenge Test and Capsaicin Inhalation Cough Challenge in a Prediction of Response to Management in Adults With a Chronic Cough.
Brief Title: MCT and Capsaicin Provocation Challenge in Diagnosis of Chronic Cough
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: BHR in chronic cough
Record Dates: First submitted 2017-11-08; First posted 2017-12-06 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cough; Cough Variant Asthma; Upper-Airway Cough Syndrome; GERD; Allergic Rhinitis
Keywords: Chronic Cough; Upper-Airway Cough Syndrome; GERD; Allergic Rhinitis; Methacholine Challenge Test; Cough Challenge; Capsaicin
MeSH Terms: conditions — Cough; Cough-Variant Asthma; upper airway cough syndrome; Gastroesophageal Reflux; Rhinitis, Allergic; Chronic Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cough variant asthma treatment — Evaluation of the treatment response to inhaled corticosteroids, long-acting beta-agonists, montelukast, prednisone.

SUMMARY:
The aim of the study is to assess the prevalence of bronchial hyperresponsiveness (BHR) in non-smoking adults with chronic cough and the prevalence of BHR in patients with upper airway cough syndrome (UACS) and gastroesophageal reflux disease (GERD), to evaluate the relationship between BHR and cough reflex sensitivity, to assess the diagnostic accuracy of methacholine challenge test (MCT) in cough variant asthma (CVA) with special regard to its discriminating cut off value between CVA and other causes of chronic cough, particularly GERD, to estimate prognostic value of BHR, fractional exhaled nitric oxide (FeNO) and induced sputum eosinophil count in predicting response to asthma treatment.

Patients diagnosed with a chronic cough will undergo the standard diagnostic work-up recommended by experts for patients with a chronic cough, including methacholine challenge test (MCT) and an at least 4-week period of causal treatment. Patients with BHR in MCT will be treated with - in first step B2-agonist and inhaled corticosteroid (ICS) for at least 4 weeks, if improvement is not significant in next steps with leukotriene receptor antagonist (LTRA) or systemic corticosteroid. A good treatment response, evaluated by visual analogue scale (VAS), Leicester Cough Questionnaire (LCQ) and cough challenge will confirm the diagnosis of the disease. A statistical analysis will consist of the frequency of BHR in a chronic cough, correlation between the results of MCT and cough reflex sensitivity in capsaicin inhalation test and cut-off point for MCT to discriminate asthma from other causes of a chronic cough.

DETAILED DESCRIPTION:
The present study has the following objectives:

1. to assess the prevalence of BHR in non-smoking adults with a chronic cough,
2. to assess the prevalence of BHR in patients with UACS and GERD,
3. to evaluate the relationship between BHR and cough reflex sensitivity,
4. to assess the diagnostic accuracy of MCT in CVA with special regard to its discriminating value between CVA and other causes of a chronic cough, particularly GERD,
5. to estimate prognostic value of BHR, fractional exhaled nitric oxide (FeNO) and induced sputum eosinophil count in predicting response to asthma treatment.

The investigated group will consist of 80 non-smoking adults (18-75 years old), who are not treated with angiotensin-converting enzyme inhibitors, with no signs of respiratory infection within six weeks prior to enrolment, with a normal chest radiograph and who are referred to the hospital due to a cough lasting at least eight weeks.

After obtaining an informed consent, the diagnostic approach of the most common causes of chronic cough will be performed: a medical history, physical examination, chest radiograph, in some cases chest computed tomography, pulmonary function tests (spirometry, fractional exhaled nitric oxide, methacholine challenge test), laboratory tests (total immunoglobulin E concentration, complete blood count), skin prick tests, induced sputum cell count, computed tomography of the paranasal sinuses and ENT consultation, 24-hour impedance with pH monitoring, videolaryngoscopy and cough challenge with capsaicin.

The cough severity will be assessed twice (on admission and after six weeks of causal treatment) using the Visual Analogue Scale (VAS), the Polish version of the Leicester Cough Questionnaire (LCQ) and the capsaicin inhalation cough challenge.

If MCT result is positive, CVA will be assumed the cause of a chronic cough and treatment with an inhaled steroid combined with a long-acting beta-agonist will be administered for at least 4 weeks. If no satisfactory response to this treatment is observed, an anti-leukotriene agent or in the next step systemic corticosteroid will be applied. Ineffective treatment with the above-mentioned medications will indicate an opportunity for a different underlying cause of BHR. The estimation the area under a ROC (receiver operating characteristic) curve will be used to determine the optimal cut-off point for the differentiation between asthma and alternate causes of a chronic cough.

It is expected to assess the frequency of bronchial hyperresponsiveness in subjects with a chronic cough, to confirm a correlation between the results of MCT and the sensitivity of cough reflex measured in capsaicin inhalation cough challenge. The investigation will probably determine a precise cut-off point for MCT which would allow discriminating asthma from other causes of a chronic cough.

ELIGIBILITY:
Inclusion Criteria:

1. Adults patients aged between 18 and 75;
2. Chronic cough lasting more than 8 weeks;
3. Non-smoking (min. 6 months);
4. Not treated with angiotensin-converting enzyme (ACE) inhibitors;
5. Not treated with:

   1. inhaled corticosteroids or systemic corticosteroids min. 4 weeks before enrolment,
   2. proton pump inhibitors min. 2 weeks before enrolment,
   3. antihistaminic drugs 1 week before enrolment;
6. With normal chest radiograph or with insignificant changes in cough pathogenesis
7. Without airway infection in previous 6 weeks.
8. Patients enrolled with informed consent.

Exclusion Criteria:

1. Patients under 18 years old and above 75 years old;
2. Smokers (actual or ex-smokers shorter than 6 weeks);
3. Therapy with corticosteroids (inhaled or systemic) for last 4 weeks, proton pump inhibitors for 2 weeks, antihistaminic drug for 1 week before enrolment;
4. Airway infection 6 weeks preceding enrolment or during study - re-attempt to enroll after 6 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-smoking patients aged 18-75, meeting inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The decrease of a cough after cough variant asthma therapy measured by Leicester Cough Questionnaire (LCQ). | at least 4 weeks of treatment
  Increase in quality of life measured with LCQ min. 1.3 points.
The decrease of a cough after cough variant asthma therapy measured by Visual Analogue Scale (VAS). | at least 4 weeks of treatment
  Reduction of cough intensity measured by VAS: Reduction min. 20 mm in VAS
The decrease of a cough after cough variant asthma therapy measured by the cough challenge. | at least 4 weeks of treatment
  Increase capsaicin concentration causing causing two/five (C2/C5) cough episode in the cough challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Lung Diseases and Allergy Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No